CLINICAL TRIAL: NCT03948477
Title: Phase II, Randomised, Double-blinded, Placebo Controlled, Crossover Trial to Assess Pantoprazole's Effectiveness as Prophylaxis Against Delayed CINV in Patients Receiving Adjuvant or Neoadjuvant Breast Cancer Chemotherapy
Brief Title: Pantoprazole Prophylaxis Against Delayed CINV for Patients Receiving Breast Cancer Chemotherapy
Acronym: PantoCIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Dr Richard Isaacs, Medical Oncologist, University of Auckland, New Zealand
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CTNZ-2017-01
Record Dates: First submitted 2019-03-28; First posted 2019-05-14 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Oncology; Breast Cancer; Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Vomiting | interventions — Pantoprazole

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomised, crossover trial, phase II, stratified by the chemotherapy regimen
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pantoprazole/Placebo (Other): Participants will take one 40 mg capsule of Pantoprazole daily for 5 days at the beginning of cycle 1 then they will take one capsule of matched Placebo daily for 5 days at the beginning of cycle 2
  Interventions: Drug: Pantoprazole 40mg; Drug: Placebo
- Placebo/Pantoprazole (Other): Participants will take one capsule of matched Placebo daily for 5 days at the beginning of cycle 1 then they will take one 40 mg capsule of Pantoprazole daily for 5 days at the beginning of cycle 2
  Interventions: Drug: Pantoprazole 40mg; Drug: Placebo

INTERVENTIONS:
Drug: Pantoprazole 40mg — Proton pump inhibitor, drug action is to irreversibly block the hydrogen-potassium adenosine triphosphatase enzyme system (the 'proton pump') of the gastric parietal cell. This reduces basal and stimulated gastric acid secretion therefore raising gastric pH.
  Other Names: Apo-Pantoprazole
Drug: Placebo — Matched placebo

SUMMARY:
This study explores whether a commonly used medication called Pantoprazole can help prevent delayed nausea and vomiting from chemotherapy for early breast cancer.

Delayed nausea, and occasionally vomiting, can occur after breast cancer chemotherapy, affecting quality of life. A potential cause of these delayed side effects is that the chemotherapy may cause stomach irritation. Pantoprazole is commonly used to treat stomach irritation by reducing stomach acid, which may in turn improve nausea and/or vomiting.

Patients undergoing breast cancer chemotherapy before or after primary surgery will be invited to participate in the study. They will be asked how much nausea or vomiting they have with and without Pantoprazole from Day 2 until 5 after they receive chemotherapy. All participants will still receive all of the usual anti-sickness medications, which are very effective in preventing sickness in the first 24 hours after treatment, but not for delayed symptoms.

Information from the study may lead to a change in practice with patients using Pantoprazole to reduce the risks of delayed nausea and vomiting.

DETAILED DESCRIPTION:
Breast Cancer is the most common cancer type in women in New Zealand and has the second highest mortality (Ministry of Health NZ) Many women with early breast cancer still receive chemotherapy, before or after surgery and delayed nausea is a particular challenge. Ensuring tolerable therapy is critical to improving outcomes, by enabling patients to complete optimal anti-cancer therapy and to improve quality of life during therapy. Despite recent advances in antiemetic regimens, recent trials showed that rates of delayed Chemotherapy-Induced Nausea and Vomiting (CINV) are is in excess of 50%, with significant impacts on quality of life during treatment. This suggests that different mechanisms than those targeted by centrally acting anti-emetics account for such symptoms. There is strong evidence that chemotherapy regimens can result in gastrointestinal mucosal injury and dyspepsia. A number of studies have shown chemotherapy-induced dyspepsia can be relieved by a proton pump inhibitor, but none have reported their use as prophylaxis for delayed CINV, which may be a linked symptom. Proton pump inhibitors are widely used in the treatment of non-malignant dyspeptic conditions and are the most potent medications at reducing gastric acid secretions. They are considered safe in short-term use and are commonly used in clinical practice in cancer patients as well as the wider population. The pharmacokinetics Pantoprazole make it the ideal PPI for this study. The experience of New Zealand Medical Oncologists is that delayed nausea is often completely resolved by the delayed use of a PPI when symptoms occur. In this study we hope to see a 30% difference in the rates of delayed nausea by using a drug which is readily available and of very low cost. This will be the first time it has been used as preventive therapy in this setting. If this benefit occurs, it would significantly improve the treatment journey and may improve compliance to anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women who are being considered for adjuvant or neoadjuvant chemotherapy with either FEC or AC or TC chemotherapy and have been deemed by their treating Oncologist as being fit for treatment. The scheduled length of each chemotherapy cycle must be 14-21 days.
2. Age ≥18 years.
3. Willing to comply with all study requirements, including treatment (being able to swallow tablets), timing and nature of required assessments.
4. All patients must be able to speak and read in English to ensure consent is informed and documentation of patient-reported outcome measures can be adhered to.
5. Signed, written informed consent.

   -

Exclusion Criteria:

1. Patients who are receiving therapy to reduce gastric acid (including proton pump Inhibitors (e.g. Omeprazole, Pantoprazole, Lansoprazole, Esomeprazole or Histamine type-2 receptor antagonists e.g. Ranitidine)) at the time of enrolment will be excluded from the trial.
2. Patients with pre-existing hypomagnesemia as defined by the reference range at the investigating sites laboratory.
3. Patients with a history of cardiac arrhythmias including atrial fibrillation or paroxysmal tachycardias.
4. Patients with known metastatic disease.
5. The presence of any serious medical or psychiatric conditions, which might limit the ability of the patient to comply with follow up.
6. The presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow up schedule, including alcohol dependence or drug abuse.
7. Pregnancy, lactation or inadequate contraception. Women must be postmenopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Reduce the incidence of delayed CINV in patients receiving adjuvant or neoadjuvant breast cancer chemotherapy | Measured on day 5, after chemotherapy
  To determine whether Pantoprazole can reduce the incidence of delayed CINV in patients receiving adjuvant or neoadjuvant breast cancer chemotherapy (as measured on day 5 using the MASCC Antiemesis Tool (MAT) to assess nausea over days 2-5 of each chemotherapy cycle) as compared to placebo. Specifically, the primary endpoint will be the complete absence of both nausea and vomiting during days 2-5.

SECONDARY OUTCOMES:
Nausea MAT scores | Days 2-5 following chemotherapy for cycle 1 and 2 (each cycle is either 14 or 21 days)
  Whether Pantoprazole improves nausea MAT scores over days 2-5
Vomiting MAT scores | Days 2-5 following chemotherapy for cycle 1 and 2 (each cycle is either 14 or 21 days)
  Whether Pantoprazole reduces the number of episodes of vomiting (MAT) over days 2-5
Heartburn improvement | Days 2-5 following chemotherapy for cycle 1 and 2 (each cycle is either 14 or 21 days)
  Whether Pantoprazole improves heartburn score (measured using the FSSG for reflux and/or dyspepsia) as self-reported on day 5 regarding days 2-5.
Heartburn and Nausea scores | Days 2-5 following chemotherapy for cycle 1 and 2 (each cycle is either 14 or 21 days), using a regression model, with allowance for a possible non-linear relationship.
  Whether FSSG scores (heartburn) are associated with the MAT nausea scores reported by the patient over days 2-5.
Use of breakthrough medications | Days 2-5 following chemotherapy for cycle 1 and 2 (each cycle is either 14 or 21 days)
  Whether Pantoprazole lowers the requirement for breakthrough medications (as self-recorded by the patients on days 2-5).
Patient preference | end of chemotherapy cycle 2 (cycle 2 is either 14 or 21 days)
  Whether Pantoprazole is preferred by patients over Placebo (by using a patient preference survey at the end of cycle 2).
Adverse events | From date of consent to 28 days after the last study treatment
  To assess whether adverse events (including hypomagnesemia, diarrhoea, abdominal pain and headache as defined by CT CAE version 4.03) are more common on Pantoprazole than on Placebo.

OTHER OUTCOMES:
Effect of chemotherapy regimen impacts use of Pantoprazole in terms of delayed CINV | Measured on day 5, after chemotherapy
  Whether the chosen chemotherapy regimen (FEC vs AC vs TC) has an impact on the benefits of Pantoprazole in terms of delayed CINV, (as measured on day 5 using the MASCC Antiemesis Tool (MAT) to assess nausea over days 2-5 of each chemotherapy cycle) as compared to placebo.
Cycle effect | Cycle 1 to end of cycle 2 (each cycle is either 14 or 21 days)
  To determine whether there is a cycle effect with respect to the incidence of delayed CINV as measured with the MAT (as measured on day 5 using the MASCC Antiemesis Tool (MAT) to assess nausea over days 2-5 of each chemotherapy cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Isaacs, MBChB FRACP, Principal Investigator — Midcentral Regional Cancer Centre Services; Navin Wewala, MBChB FRACP, Principal Investigator — Midcentral Regional Cancer Centre Services
Locations (10):
- New Zealand (10):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Taranaki Base Hospital, New Plymouth
  - Palmerston North Hospital, Palmerston North
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
  - Whangarei Hospital, Whangarei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wewala N, Kim Y, Sharples K, Benge S, Cartwright R, Tan A, Clement L, Huang Y, Wilson S, Kuper-Hommel M, Barton S, Jones J, Bremer L, Hari Dass P, Wrigley A, Findlay M, Isaacs R. Proton pump inhibition to prevent delayed chemotherapy-induced nausea and vomiting in patients receiving adjuvant or neoadjuvant breast cancer chemotherapy: a phase II, randomised double-blind crossover trial (PantoCIN). Support Care Cancer. 2025 May 20;33(6):484. doi: 10.1007/s00520-025-09528-0. PMID 40394328
- See also: Cancer Trials New Zealand website study record — http://cancertrialsnz.blogs.auckland.ac.nz/pantocin
- See also: Breast Cancer Foundation website study record (Co-funder) — https://www.breastcancerfoundation.org.nz/clinical-trials/clinical-trial/pantocin-